CLINICAL TRIAL: NCT05544747
Title: Comparison of Action Observation Therapy Versus Mirror Therapy on Upper Limb Physical Performance and Quality of Life in Stroke
Brief Title: Action Observation Therapy Versus Mirror Therapy on Upper Limb in Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-01332 Sania
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy (Experimental): The patients in the action observation therapy group will be required to observe the upper limb movements or functional actions in video clips. (i.e., the observation phase) and to execute what they had observed to the best of their ability (i.e., the execution phase). Three common categories of movements and tasks will be elected in the action observation therapy protocol based on the related literature
  Interventions: Other: Action Observation Therapy
- Mirror Therapy (Active Comparator): During the mirror therapy, the patients will be seated in front of a mirror box placed at their mid-sagittal plane. The affected arm of the participants will be placed inside the mirror box and the unaffected arm in front of the mirror. The patient will be instructed to watch the mirror reflection of the movement performed by his/her unaffected hand carefully and to imagine that the movement was performed by the affected hand.
  Interventions: Other: Mirror Therapy

INTERVENTIONS:
Other: Action Observation Therapy — following phases will be included in action observation therapy group:
  1. upper limb active range of motion (AROM) exercises.
  2. reaching movement or object manipulation.
  3. upper limb functional tasks.
  Arms: Action Observation Therapy
Other: Mirror Therapy — following phases will be included in mirror therapy group:
  1. AROM exercises),
  2. reaching movement or object manipulation, and
  3. functional task practice
  Arms: Mirror Therapy

SUMMARY:
Stroke is a medical condition which causes the cessation of blood flow to the brain cells and results in cell death and ultimately can lead to motor disorders, perception disorders, language disorders, sensory disturbances.It is well known that stroke is the leading cause of death and one of the greatest causes of long-term motor disability in adults.The incidence of stroke is increasing day by day in low-income countries as compared to high-income countries because of the effects of not using evidence-based practice in health-related conditions in low-income countries. In the last few years, several approaches have been used for the recovery of hand dexterity after stroke. Among them, the Mirror therapy, task-oriented therapy, robot-assisted rehabilitation and action observation has gained greatest attention.Action observation training is one of the new developing rehabilitation technique that targets motor learning by the activation of mirror neurons and is the most important approach that targets the motor and functional recovery in stroke patients. In action observation training, the movements are produced because of the external stimuli in which actually the visual attention recruit the cerebellar-thalamic-cortical circuit of the brain. Action observation is based on activities of the motor neuron system and they discharge mostly in association with complex tasks as compared to simple tasks.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Middle cerebral artery stroke
* 1 to 6 months of stroke onset
* Baseline score of the Fugyl Myer Assessment is between 20 and 60 for the upper limb.
* Modified Ashworth scale with a score of 2 Ability to follow the study instructions-Mini mental state examination (MMSE) score >25

Exclusion Criteria:

* Participants failing to fall in this category would be excluded from the study.
* Patients who cannot perform the active movement of the upper limb in pre-stroke condition due to musculoskeletal problems
* cardiopulmonary diseases which could hinder their ability to participate in the rehabilitation program in this study
* Patient with impaired cognition

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Fugel Meyer assessment scale for upper limb | week 6
  An assessment scale for post stroke hemiplegic patients and is performance-based impairment index. This scale is having 5 domains namely Motor functioning, Sensory Functioning, Balance, Joint Range of Motion and Joint pain. I divided the motor functioning for upper extremity into 0 to 66 points and evaluates mobility, speed and coordination
Box and Block Test (BBT) | week 6
  This test is used to evaluate the manual dexterity of post stroke patients. BBT is composed of wooden box with two equal compartments having 150 boxes in one compartment and patient is asked to move the boxes from one compartment to another within 60 seconds. Before starting the test an extra 15 seconds time is given to the patient for familiarization with the test. First the patient performed the activity with the healthy arm and then with the affected arm. Scoring is done on the basis of the number of boxes transferred from one compartment to another within 60 seconds
Functional Independence Measure (FIM) | week 6
  The FIM is a commonly used scale for assessing the performance in basic daily activities. It contains 18 items (i.e., 13 motor and 5 cognition items), and the total score ranges from 0 to 126

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) version 3.0 | week 6
  The SIS 3.0 is a stroke-specific, patient-reported questionnaire for evaluating the function, participation, and health-related quality of life of stroke survivors. The SIS 3.0 has sound psychometric properties. It consists of 59 items, and higher scores indicate better function and greater participation.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Helping hand institute of rehabilitation sciences, Mansehra, Pakistan

IPD SHARING:
Plan to Share IPD: No